CLINICAL TRIAL: NCT06014788
Title: NPWTi vs. Conventional NPWT in Superficial and Deep Abdominal Surgical Site Infections
Brief Title: Is the NPWTi Better Than the Conventional NPWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Medical Academy, Bulgaria (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20.08.1964
Record Dates: First submitted 2023-07-28; First posted 2023-08-28 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Wound Infection Superficial Incisional; Postoperative Wound Infection Deep Incisional Surgical Site
Keywords: NPWTi; conventional NPWT; superficial and deep SSIs

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPWTi (Experimental): The whole wound was filled with black foam (Granufoam®, KCI). The instillation was performed via gravity from i.v. bag through a drain put within the foam. Chlorhexidine 0.1% 300 ml in 700 ml saline was used for continuous instillation three times daily (3 L per day) on the background of continuous pressure of 125 mmHg. The dressing changes were performed every 48-72 hours.
  Interventions: Device: NPWTi
- conventional NPWT (Active Comparator): The wound was filled with black foam (Granufoam®, KCI) and covered with plastic folio. A continuous pressure of 125 mmHg was applied using the hospital suction system. The dressing changes were performed every 48 hours.
  Interventions: Device: Conventional NPWT

INTERVENTIONS:
Device: NPWTi — The wound was filled with black foam (Granufoam®, KCI). The instillation was performed via gravity from i.v. bag through a drain put within the foam. Chlorhexidine 0.1% 300 ml in 700 ml saline was used for continuous instillation three times daily (3 L per day) on the background of continuous pressure of 125 mmHg.
  Arms: NPWTi
Device: Conventional NPWT — Conventional NPWT
  Arms: conventional NPWT

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of NPWTi and NPWT in superficial and deep surgical site infections using an improvised system with continuous lavage with saline and chlorhexidine. The main question it aims to answer is whether the NPWTi is better than conventional NPWT. Participants will be given NPWTi or conventional NPWT.

Researchers will compare the two groups to see if NPWTi diminishes the rate of recurrent infections and the number of reoperations, shortens the hospital stay, and alleviates the burden on the hospital staff in comparison to the conventional NPWT.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years
* superficial or deep SSIs after laparotomy or laparoscopic surgery

Exclusion Criteria:

* persons < 18 years
* documented inherited or acquired coagulation disorders or platelet deficiency
* presence of deep space infection (intra-abdominal abscess or ongoing peritonitis)
* prosthetic material infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
eradication of the infection | 6 weeks
  (negative microbiology or bacterial count < 103)
the rate of wound closure | 6 weeks
  the wound closure by suture or flap
30-day recurrence rate | 30 days after discharge
  30-day recurrence rate of the infection

SECONDARY OUTCOMES:
hospital stay | 6 weeks
  hospital stay in days
number of OR visits | 6 weeks
  number of OR visits and dressing changes under general anesthesia
time to wound closure | 6 weeks
  the time elapsed from the start of the treatment to wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Ventsislav Mutafchiyski, DSc, FACS, Principal Investigator — Military Medical Academy, Bulgaria
Locations (1):
- Department of Sugery, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No